CLINICAL TRIAL: NCT02106715
Title: Overuse Injuries in Road Cyclists, Prevalence and Prevention
Acronym: Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Joanna Kvist, Associate Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cycle_Dnr2014/42-31
Record Dates: First submitted 2014-03-23; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Overuse Injuries
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Active Comparator): Two exercises for training of core stability and mobility.
  Interventions: Other: Training
- Control (No Intervention): Control group without training

INTERVENTIONS:
Other: Training — Two exercises for training of core stability and mobility.
  Arms: Training

SUMMARY:
The purpose of this study is to investigate the prevalence of overload injuries to road cyclists in Sweden, and if it 's possible to prevent low back pain by a simple exercise program for two months of training .

ELIGIBILITY:
Inclusion Criteria:

* Planning to ride "Vätternrundan 2014" in a subgroup .
* Cycled "Vätternrundan" at least twice in the past or bicycled for exercise at least 800 mil ( the equivalent of two seasons) .
* Age 18-55 years .
* Training cycle at least three hours a week or three days a week .

Exclusion Criteria:

* Do not have access to a computer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number and type of overuse injuries | Four months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Div Physiotherapy, Linkoping University, Linköping, Sweden

REFERENCES:
- [Derived] Garrosa-Martin G, Muniesa CA, Molina-Martin JJ, Diez-Vega I. Low Back Pain in Cycling. Are There Differences between Road and Mountain Biking? Int J Environ Res Public Health. 2023 Feb 21;20(5):3791. doi: 10.3390/ijerph20053791. PMID 36900802